CLINICAL TRIAL: NCT00428441
Title: The Negative Predictive Value of D-dimer on the Risk of Recurrent Venous Thromboembolism in Patients With Multiple Previous Events: a Prospective Cohort Study
Brief Title: D-dimer to Predict Recurrence in Patients With Multiple Episodes of Venous Thromboembolism
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrolment was halted prematurely because of the observed excess in recurrences
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Walter Ageno, Associate Professor of Internal Medicine, Università degli Studi dell'Insubria
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2175
Record Dates: First submitted 2007-01-26; First posted 2007-01-30 (Estimated); Results first posted 2011-09-26 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-08

CONDITIONS: Venous Thromboembolism
Keywords: D-dimer; Recurrence; Venous thromboembolism
MeSH Terms: conditions — Venous Thromboembolism; Recurrence | interventions — Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Warfarin — tablets, based on INR levels, according to D-dimer levels

SUMMARY:
Optimal duration of oral anticoagulant therapy in patients with recurrent episodes of venous thromboembolism (VTE) is a matter of debate and recommendations are based on inadequate evidence. More than 12 months of treatment are currently recommended, and the grade of recommendation is low.

The PROLONG study has recently evaluated the predictive role of D-dimer measurement after withholding oral anticoagulant treatment in patients with a first episode of VTE. Patients with a positive D-dimer had a significantly higher incidence of VTE recurrences than patients with a negative D-dimer and required resumption of the antithrombotic treatment. Based on the results of this and of previous cohort studies, it appears safe to withhold treatment in patients with negative D-dimer values and to continue treatment in patients with altered D-dimer levels.

Aim of this study is therefore to assess the negative predictive value of D-dimer also in patients with recurrent VTE and to evaluate the clinical utility of this approach in this patient setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least two episodes of objectively documented venous thromboembolism (at least one proximal deep vein thrombosis or pulmonary embolism)
* Ongoing treatment with oral anticoagulants for at least a) 12 months in case idiopathic DVT was the last event; b) 6 months in all other cases
* Age > 18 years
* Informed consent provided

Exclusion Criteria:

* Pregnancy/puerperium
* One or more episodes of massive pulmonary embolism
* Last event isolated idiopathic pulmonary embolism
* Two or more idiopathic VTE events
* First degree relatives with recurrent VTE
* Right ventricular disfunction or pulmonary hypertension
* Active cancer
* Antiphospholipid antibodies syndrome
* Antithrombin deficiency
* Homozygous Factor V Leiden or G20210A prothrombin mutation
* Heterozygous Factor V Leiden and G20210A prothrombin mutation
* Concomitant congenital thrombophilic mutations
* Concomitant indications to long term oral anticoagulant treatment
* Severe cardiorespiratory insufficiency
* Severe liver or renal disease (creatinine clearance > 2 mg/dL)
* Limited life expectancy
* Geographic inaccessibility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2007-05; Primary Completion 2010-06 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gualtiero Palareti, Study Chair — University of Bologna; Walter Ageno, Study Director — Università degli Studi dell'Insubria; Vittorio Pengo, Study Director — University of Padova
Locations (1):
- University Of Insubria, Varese, Italy

REFERENCES:
- [Background] Palareti G, Cosmi B, Legnani C, Tosetto A, Brusi C, Iorio A, Pengo V, Ghirarduzzi A, Pattacini C, Testa S, Lensing AW, Tripodi A; PROLONG Investigators. D-dimer testing to determine the duration of anticoagulation therapy. N Engl J Med. 2006 Oct 26;355(17):1780-9. doi: 10.1056/NEJMoa054444. PMID 17065639
- [Background] Palareti G, Legnani C, Cosmi B, Guazzaloca G, Pancani C, Coccheri S. Risk of venous thromboembolism recurrence: high negative predictive value of D-dimer performed after oral anticoagulation is stopped. Thromb Haemost. 2002 Jan;87(1):7-12. PMID 11848459

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment period 2007-2009 location Thrombosis centers
Groups:
- D-dimer Negative: patients with recurrent venous thrombosis and negative D-dimer at the time of enrolment
Period: Overall Study
Arm/Group | D-dimer Negative
Started | 75
Completed | 74
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | D-dimer Negative
Number analyzed (Participants) | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 43
  >=65 years | 32
Age Continuous [Mean (Standard Deviation); unit: years] | 61.9 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 41
Region of Enrollment [Number; unit: participants]
  Italy | 75

OUTCOME MEASURES:

1. Primary Outcome: Recurrent Deep Vein Thrombosis or Pulmonary Embolism in Patients With Persistently Negative D-dimer Levels
Description: Objectively documented deep vein thrombosis, pulmonary embolism, superficial vein thrombosis
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | D-dimer Negative
Number analyzed (Participants) | 75
participants | 9

2. Primary Outcome: Rate of Patients With Altered D-dimer Levels and Temporal Distribution of Alterations
Time Frame: 3 months
Reporting Status: Not Posted

3. Secondary Outcome: Recurrent Deep Vein Thrombosis or Pulmonary Embolism in Patients Who Resumed Oral Anticoagulant Therapy
Time Frame: 3 months
Reporting Status: Not Posted

4. Secondary Outcome: Incidence of Major Bleeding in Patients Who Resumed Oral Anticoagulant Therapy
Time Frame: 3 months
Reporting Status: Not Posted

5. Secondary Outcome: Mortality
Time Frame: 3 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | D-dimer Negative
Serious Adverse Events (participants affected / at risk) | 0/75
Other Adverse Events (participants affected / at risk) | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No